CLINICAL TRIAL: NCT03164070
Title: Study of the Laboratory-based Evaluation of the Degrees of Activity of Medium and Large Joint Osteoarthritis
Brief Title: Study of the Laboratory-based Evaluation of the Degrees of Activity of Osteoarthritis
Status: Completed | Type: Observational
Sponsor: The Republican Research and Practical Center for Epidemiology and Microbiology (Other)
Collaborators: Belarusian Medical Academy of Post-Graduate Education (Other)
Responsible Party: Principal Investigator, Andrei Y. Hancharou, Head of the Laboratory for Immunology and Cellular Biotechnology, The Republican Research and Practical Center for Epidemiology and Microbiology
Other Study IDs: RRPCEM_OA
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Flow cytometry; Synovial fluid
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Synovial fluid samples stored in the tube with sodium heparin. Venous blood samples drained into tube with sodium heparin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with osteoarthritis: Patients with medium and large joint osteoarthritis
- Control group: Control group of healthy persons

SUMMARY:
This study evaluates laboratory-based method to estimate the degrees of activity of medium and large joint osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a chronic progressive disease, characterized by degradation of joint cartilage, synovial inflammation and joint dysfunction. This study evaluates laboratory-based method to estimate the degrees of activity of medium and large joint OA. Samples of synovial fluid (SF) from the patients with the OA (ICD-10 codes: M15, M16 and M17) will be assessed for T-cell subsets, msast cells, fibroblast-like synoviocytes (FLS) and macrophage-like synoviocytes (MLS) by flow cytometry. Subpopulations of blood T-cells involved in the inflammation will also be assayed. Standard clinical investigation will be performed and the results will be used to estimate the laboratory criteria or degrees of activity of medium and large joint OA.

ELIGIBILITY:
Inclusion Criteria:

* medium and large joint active osteoarthritis

Exclusion Criteria:

* refuse of patient to participate in the trial;
* acute infectious diseases;
* pregnancy/lactation;
* intercurrent severe chronic diseases;
* HIV, Hepatites B/C;
* active tuberculosis;
* alcohol use disorder/drug addiction;
* malignant neoplasms/leukemia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with medium and large joint osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
The sensitivity of the proposed laboratory-based method in the diagnostics of the activity of osteoarthritis | 2 month
  The sensitivity of the proposed laboratory-based method in the diagnostics of the activity of medium and large joint osteoarthritis

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Y Hancharou, Dr, Study Director — Head of the Laboratory for Immunology and Cellular Biotechnology, The Republican Research and Practical Center for Epidemiology and Microbiology
Locations (1):
- Andrei Hancharou, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No